CLINICAL TRIAL: NCT04445597
Title: ANalyzing Olfactory Dysfunction Mechanisms In COVID-19
Acronym: ANOSMIC-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Max Planck Research Unit for Neurogenetics (Unknown); AZ Sint-Lucas Brugge (Other); Universitair Ziekenhuis Brussel (Other); Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Laura Van Gerven, Professor doctor, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S64042
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: SARS-CoV-2
Keywords: Hyposmia; Anosmia; Olfactory Dysfunction; COVID-19; SARS-CoV-2
MeSH Terms: conditions — Anosmia; COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COVID-19 positive or negative patients (Other): Hospitalised patients with or without COVID-19 (with or without olfactory dysfunctions)
  Interventions: Other: Sampling of tissue

INTERVENTIONS:
Other: Sampling of tissue — In all groups of participants, tissue from the nasal cavity and olfactory system will be surgically removed

SUMMARY:
We aim to understand the mechanism of olfactory dysfunction in COVID-19.

DETAILED DESCRIPTION:
In December 2019, a new coronavirus causing severe acute respiratory syndrome was described in Wuhan, China. This virus, later named severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), spread worldwide and has been designated a pandemic by the World Health Organization.

By the beginning of March 2020, several Ear, Nose, Throat societies raised awareness of a frequent association between coronavirus disease 2019 (COVID-19) and smell disorders.

In the present study, the investigators wish to begin to understand the pathogenesis of olfactory dysfunction in COVID-19.

ELIGIBILITY:
Inclusion Criteria:

- Deceased hospitalised patients, tested positive or negative for SARS-CoV-2 for patient or control group respectively

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-05-07 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of SARS-CoV-2 in the sampled tissue | Immediately after death
  In the sampled tissues, the investigators will determine presence of SARS-CoV-2 by means of immunohistochemistry, RNA-scope and spatial transcriptomics

CONTACTS AND LOCATIONS:
Overall Officials: Laura Van Gerven, Principal Investigator — UZ/KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No